CLINICAL TRIAL: NCT01206868
Title: Prospective Open Randomized Study to Evaluate the Efficiency of Prophylactic Fenestration of the Peritoneum in Kidney Transplantation in Preventing the Occurrence of Postoperative Lymphoceles
Brief Title: Prophylactic Fenestration of the Peritoneum in Kidney Transplantation
Acronym: PROFFEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Tim Scholz MD, PhD. Principal Investigator, Section for Transplant Surgery, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S-06342a
Record Dates: First submitted 2010-09-21; First posted 2010-09-22 (Estimated); Last update posted 2010-09-22 (Estimated); Status verified 2007-03

CONDITIONS: Incidence of Symptomatic Lymphocele After Kidney Transplantation; Prevalence of Perirenal Fluid Collections at One, Five and Ten Weeks
Keywords: kidney, transplantation, surgery, complications, lymphocele, fluid collections.
MeSH Terms: conditions — Lymphocele | interventions — Fenestration, Labyrinth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fenestration (Active Comparator): Fenestration of the peritoneum according to the length of the transplanted kidney
  Interventions: Procedure: Fenestration
- Control (Sham Comparator): Standard kidney transplantation
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: Fenestration — Fenestration of the peritoneum according to the length of the transplanted kidney
  Arms: Fenestration
Procedure: Control — Standard kidney transplantation
  Arms: Control

SUMMARY:
A single centre open randomised parallel-group study to evaluate whether prophylactic fenestration of the peritoneum at the time of renal transplantation prevents lymphocele formation.

Adult (>18 years old) recipients of renal transplants from deceased donors were eligible for inclusion. From March 2007 to May 2009 130 patients were included. The patients were randomized either to peroperative peritoneal fenestration, or to serve as controls. Block-randomization was conducted in groups of 10, drawn from envelopes containing five notes from each group. Patients who previously had undergone extensive abdominal surgery, or were included in other studies were excluded.

ELIGIBILITY:
Inclusion Criteria:

* Adult recipients of kidney transplants from deceased donors

Exclusion Criteria:

* Former extensive abdominal surgery
* Participation in other studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2007-03; Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Incidence of symptomatic lymphoceles | 1 - 3 years
  Symptomatic lymphoceles treated by surgical intervetion or ultrasound guided drainage

SECONDARY OUTCOMES:
Prevalence of fluid perirenal collections evaluated by ultrasound at 1, 5 and 10 weeks | 1 -10 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Oslo, Norway

REFERENCES:
- [Derived] Syversveen T, Midtvedt K, Brabrand K, Oyen O, Foss A, Scholz T. Prophylactic peritoneal fenestration to prevent morbidity after kidney transplantation: a randomized study. Transplantation. 2011 Jul 27;92(2):196-202. doi: 10.1097/TP.0b013e318220f57b. PMID 21597401